CLINICAL TRIAL: NCT01832337
Title: Limb Remote Ischemic Preconditioning for Heart and Intestinal Protection During Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fei Li (Other)
Responsible Party: Sponsor-Investigator, Fei Li, Sixth Affiliated Hospital, Sun Yat-sen University, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 伦研批第E201215号
Record Dates: First submitted 2013-03-16; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Laparoscopic Colorectal Surgery

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- precondition (Experimental)
  Interventions: Procedure: Limb remote ischemic preconditioning (LRIP)

INTERVENTIONS:
Procedure: Limb remote ischemic preconditioning (LRIP) — Limb remote ischemic preconditioning (LRIP) consisted of three cycles of left upper limb ischemia induced by inflating a blood pressure cuff on the left upper arm to 200mmHg, with an intervening 5 minutes of reperfusion, during which time the cuff was deflated.

SUMMARY:
Remote ischaemic preconditioning may confer the cytoprotection in critical organs. The investigators hypothesized that limb remote ischemic preconditioning (RIPC) would reduce heart and gastrointestinal function injury in middle-aged and elderly patients undergoing elective laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* age >40 years old
* ASA I-II
* receive elective laparoscopic colorectal surgery
* written informed consent can be obtained

Exclusion Criteria:

* coagulation disorders
* patients with cardiac pacemaker
* patients with severe cardiac,or pulmonary,hepatic,renal disease ,or can not tolerate laparoscopic surgery
* patients with peripheral vascular disease affecting the upper limbs
* patients with mental,or hearing, vision disorder, who is not able to communicate with physicians
* difficult airways that can not receive rapid induction

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Limb remote ischemic preconditioning may have effective protection of heart and intestinal in middle-aged and elderly patients undergoing elective laparoscopic colorectal surgery. | within the first 7 days after surgery
  We hypothesized that limb remote ischemic preconditioning (RIPC) would reduce heart and intestinal injury in patients undergoing elective laparoscopic colorectal surgery.The primary outcomes included the biomarkers reflecting intestinal injury (serum intestinal fatty acid binding protein, endotoxin levels and),time (hours) from end of operation to first passage of stool or flatus,the biomarker reflecting heart injury (CTnI,serum heart fatty acid binding protein ).Perioperative electrocardiographic was also recorded. In addition, the severity of intestinal injury was assessed with pathological scoring methods. Markers of systemic inflammation (CRP) were measured as well.

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China